CLINICAL TRIAL: NCT05552144
Title: Exploring Caregivers' Experiences Related to the Use of a Smart Toothbrush by Children With Autism Spectrum Disorder
Brief Title: Documenting Toothbrushing Experiences of Caregivers Who Care for Children With Autism Spectrum Disorders
Acronym: humBrush
Status: Completed | Type: Observational
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Other Study IDs: 850364
Record Dates: First submitted 2022-07-21; First posted 2022-09-23 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: ASD I; ASD2
Keywords: autism spectrum disorder; ASD; Smart toothbrush; Caregiver experience
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Hum by Colgate Smart Kids Toothbrush (battery powered) - 490000006871 — The first 15 caregivers and their children who meet the inclusion/exclusion characteristics and sign an Informed Consent Form/provide assent will be entered into the study. The caregivers will be asked to supervise the tooth brushing experience of the children with hum Kids toothbrush twice a day for 4 weeks using the associated app. The caregivers will also be asked to fill out questionnaires and participate in interviews regarding the children's brushing habits and experiences.
  Other Names: Hum by Colgate Smart Manual Kids Toothbrush - 461000001191 (toothbrush), 461000001968 (MAGIK attachment)

SUMMARY:
The objective of this study is to examine caregiver reactions to the use of the hum by Colgate Smart Kids Toothbrush and associated app by children with autism spectrum disorder (ASD).

DETAILED DESCRIPTION:
This is a single-center, pretest-posttest, non-randomized, clinical study involving interviews with caregivers prior to utilization of the research toothbrush and after 4 weeks of product use by the child. All participants enrolled will be children ages 5-12 years and their primary caregivers. Participants will be asked to utilize a Hum by Colgate Smart Kids Toothbrush (manual or battery-powered) for four weeks.

To assure that subjects are comfortable with the oral care regime proposed, toothbrushes will be distributed based on the subject's previous oral hygiene habits. Children who are currently using manual brushes will receive the Hum by Colgate Smart Manual Kids Toothbrush, likewise, children who are used to battery-powered toothbrushes will receive the Hum by Colgate Smart Kids battery-powered toothbrush.

All the participants will be offered the electric toothbrush and will have a chance to try it during the first visit.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form by the child's legal guardian on behalf of the child and from the primary (responsible for child's oral healthcare) caregiver.
2. Caregiver must be able to observe the child using the Hum by Colgate Smart Manual Kids Toothbrush and app twice a day.
3. Caregivers must have a child between the ages of 5-12 years old, who is willing to participate.
4. Child must be reported in good general health and good oral health based on the opinion of the study investigator.
5. Caregiver and child must be available for the duration of the study.
6. Caregiver must have access to Apple iPhone (newer than 8) or iPad (newer than 5th generation) or Android users (running Android 6.0 and up) with access to an Internet Connection.
7. Caregiver must be willing to comply with the study protocol.
8. Caregiver must be willing to download and use app associated with the connected brush.
9. Caregiver must be willing to be audiotaped during key informant interview sessions.
10. English fluency for the child's legal guardian/caregiver.
11. Caregiver must be willing to have a shared brushing experience between themselves and the child.
12. Caregiver's child must be diagnosed with ASD Level I or ASD Level II .

    1. ASD Level I: Requiring support
    2. ASD Level II: Requiring substantial support

Exclusion Criteria:

1. Child undergoing active orthodontic treatment with fixed appliances.
2. Child has obvious signs of oral disease, severe dental caries, or pain as determined by the investigator's judgment.
3. Concurrent participation by child in another clinical study.
4. Child's behavior precludes participation in the study at the investigator's discretion.
5. Current or previous use of the Hum by Colgate Smart Kids Toothbrush by the child.

Ages: 5 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: 1. 15 children, aged 5-12 years old, male and female with ASD Level I or ASD Level II.
     1. ASD Level I requires support
     2. ASD Level II requires substantial support
  2. Primary caregivers of the children.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
User experiences of hum connected toothbrush as observed by the caregiver with interviews & questionnaires. | 4 weeks
  The hum Smart Kids Toothbrush aims to capture the reactions of the caregivers of the children with ASD on the ease and usefulness of the toothbrush and the app.
  The goal is to gauge if the experience of using the connected toothbrush is ultimately enjoyable for the caregivers of the children with ASD.
  Insights from the caregivers will assist in exploring the value of utilizing "smart" toothbrush technologies for oral hygiene in children with ASD.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine France, DMD, MBE, Principal Investigator — Penn Dental School of Medicine
Locations (1):
- Penn Dental School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
All information may be stored or shared for future research purposes. All the information will be de-identified. All audio recordings will be transcribed and de-identified. De-identified means that all identifiers have been removed. The information could be stored and shared for future research in this de-identified fashion. The information may be shared with other researchers within Penn, or other research institutions, as well as pharmaceutical, device, or biotechnology companies. It would not be possible for future researchers to identify the subjects as we would not share any identifiable information about the subjects with future researchers. This can be done without again seeking their consent in the future, as permitted by law. The future use of the information only applies to the information collected on this study.

REFERENCES:
- [Result] Como DH, Stein Duker LI, Polido JC, Cermak SA. Oral Health and Autism Spectrum Disorders: A Unique Collaboration between Dentistry and Occupational Therapy. Int J Environ Res Public Health. 2020 Dec 27;18(1):135. doi: 10.3390/ijerph18010135. PMID 33375475
- See also: Oral Health and Autism Spectrum Disorders: A Unique Collaboration between Dentistry and Occupational Therapy — https://pubmed.ncbi.nlm.nih.gov/33375475/